CLINICAL TRIAL: NCT03355469
Title: Exercise Dose and Metformin for Vascular Health in Adults With Metabolic Syndrome
Brief Title: Exercise Dose and Metformin for Vascular Health in Metabolic Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven K Malin, PhD, Principal Investigator, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19364; 1R01HL130296-01A1 (NIH); NCT04817787 (obsolete NCT alias)
Record Dates: First submitted 2017-11-07; First posted 2017-11-28 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Metformin; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Each subject will be randomly assigned to receive low intensity exercise training + placebo, high intensity exercise training + placebo, or these exercise programs with metformin.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- LoEx with Placebo (Placebo Comparator): Low intensity exercise with placebo.
  Interventions: Drug: Placebo; Behavioral: Low Intensity Exercise
- HiEx with Placebo (Placebo Comparator): High intensity exercise with placebo.
  Interventions: Drug: Placebo; Behavioral: High Intensity Exercise
- LoEx with Metformin (Active Comparator): Low intensity exercise with metformin.
  Interventions: Drug: Metformin; Behavioral: Low Intensity Exercise
- HiEx with Metformin (Active Comparator): High intensity exercise with metformin.
  Interventions: Drug: Metformin; Behavioral: High Intensity Exercise

INTERVENTIONS:
Drug: Metformin — Oral metformin 2000 mg/d for 16 weeks. Metformin dosage will follow 500 mg/d ramp up progression: Week 1 = 500 mg/d; Week 2 = 1,000 mg/d; Week 3 = 1500 mg/d; Week 4-16 = 2000 mg/d.
  Arms: HiEx with Metformin; LoEx with Metformin
Drug: Placebo — Oral placebo for 16 weeks. Placebo tablets will follow a four-stage progression: Week 1 = 1 tablet; Week 2 = 2 tablets; Week 3 = 3 tablets; Week 4-16 = 4 tablets.
  Arms: HiEx with Placebo; LoEx with Placebo
Behavioral: Low Intensity Exercise — Low intensity exercise will consist of 16 weeks of walking at ~55% of each participant's predetermined VO2max and monitored via heart rate. Supervised exercised will occur on a treadmill 3d/wk and the duration will be determined based on individual fitness levels to expand 400 kcals. Supervised exercise training will follow a three-phase progression: Weeks 1-2 = 3 supervised sessions at 75% duration; Week 3-4 = 3 supervised sessions at 87% duration; Weeks 5-16 = 3 supervised sessions at 100% duration. Unsupervised exercised will be 2d/wk and the duration will half the time of the supervised training sessions.
  Other Names: LoEx
  Arms: LoEx with Metformin; LoEx with Placebo
Behavioral: High Intensity Exercise — High intensity exercise will consist of 16 weeks of walking at ~85% of each participant's predetermined VO2max and monitored via heart rate. Supervised exercised will occur on a treadmill 3d/wk and the duration will be determined based on individual fitness levels to expand 400 kcals. Supervised exercise training will follow a three-phase progression: Weeks 1-2 = 3 supervised sessions at 75% duration; Week 3-4 = 3 supervised sessions at 87% duration; Weeks 5-16 = 3 supervised sessions at 100% duration. Unsupervised exercised will be 2d/wk and the duration will half the time of the supervised training sessions.
  Other Names: HiEx
  Arms: HiEx with Metformin; HiEx with Placebo

SUMMARY:
Health organizations recommend exercise in an intensity based manner to promote cardiovascular adaptation and prevent disease. Metformin is a common anti-diabetes medication that reduces future type 2 diabetes and cardiovascular disease (CVD) risk. However, the optimal dose of exercise to be combined with metformin for vascular health remains unknown. The purpose of this study is to evaluate whether combining high or low intensity exercise with metformin has the potential to outperform either exercise intensity alone on blood flow across the arterial tree as well as impact insulin action in individuals with metabolic syndrome. Identification of such outcomes will indicate 1) whether and how metformin should be combined with physical activity for CVD prevention, 2) provide the first indication of whether exercise intensity reduces CVD risk via multi-level vasculature function vs. metabolic insulin action, and 3) provide a rational early treatment for people with metabolic syndrome to prevent/treat type 2 diabetes and CVD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 and ≤80 years old.
* Has a body mass index ≥25 and ≤47 kg/m2.
* Not diagnosed with Type 2 or Type 1 diabetes
* Not currently engaged in > 150 min/wk of exercise
* Weight stable (<2kg weight change in past 3 months)
* Non-smoking >5 years

At minimum, subject will have abdominal obesity (increased waist circumference as defined below) and may have any additional National Cholesterol Education Adult Treatment Panel III Metabolic Syndrome criteria:

* Increased waist circumference (≥102 cm in men; ≥88 cm in women)
* Elevated triglycerides (≥150 mg/dl), or on medication for treating the condition
* Reduced HDL-cholesterol (<40mg/dl in men, <50 mg/dl in women), or on medication for treating the condition
* High blood pressure (≥130 mmHg systolic or ≥85mmHg diastolic), or on medication for treating the condition
* Elevated fasting glucose (≥100 mg/dl), or on medication for treating the condition
* Other major risk factors to be noted based on the Framingham Risk Score
* HbA1c 5.7-6.4%
* LDL > 130 mg/dL
* Family history of type 2 diabetes (immediate family, i.e. parent/sibling)
* History of gestational diabetes
* History of Polycystic Ovarian Syndrome
* Family history of pre-mature cardiovascular disease (immediate family i.e. parent/sibling) before 55 for males or 65 for females that can include heart attack, peripheral arterial disease, abdominal aortic aneurysm, symptomatic carotid artery disease or clinical coronary heart disease)
* Age ( > 45 years old for men; > 55 years old for women)
* Black/African American, Mexican, Asian, and/or Hispanic
* Subjects currently taking medications that affect heart rate and rhythm (i.e. Ca++ channel blockers, nitrates, alpha- or beta-blockers)

Exclusion Criteria:

* Subjects prescribed metformin or have taken metformin within 1 year.
* Subjects with abnormal estimated glomerular filtration rate (eGFR).
* Hypertriglyceridemic (>400 mg/dl) and hypercholesterolemic (>260 mg/dl) subjects
* Hypertensive (>160/100 mmHg)
* Subjects with a history of significant metabolic, cardiac, congestive heart failure, cerebrovascular, hematological, pulmonary, gastrointestinal, liver, renal, or endocrine disease or cancer that in the investigator's opinion would interfere with or alter the outcome measures, or impact subject safety.
* Pregnant (as evidenced by positive pregnancy test) or nursing women
* Subjects with contraindications to participation in an exercise training program
* Currently taking active weight suppression medication (e.g. phentermine,orlistat, lorcaserin, naltrexone-bupropion in combination, liraglutide, benzphetamine, diethylpropion, phendimetrazine)
* Known hypersensitivity to perflutren (contained in Definity)
* Subjects who are considered non-English speaking individuals

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Malin, PhD, Principal Investigator — Rutgers University - New Brunswick
Locations (1):
- Rutgers University Loree Gymnasium, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laurent S, Katsahian S, Fassot C, Tropeano AI, Gautier I, Laloux B, Boutouyrie P. Aortic stiffness is an independent predictor of fatal stroke in essential hypertension. Stroke. 2003 May;34(5):1203-6. doi: 10.1161/01.STR.0000065428.03209.64. Epub 2003 Apr 3. PMID 12677025
- [Background] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Fernando Costa. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute scientific statement: Executive Summary. Crit Pathw Cardiol. 2005 Dec;4(4):198-203. doi: 10.1097/00132577-200512000-00018. No abstract available. PMID 18340209
- [Background] DeFronzo RA, Abdul-Ghani M. Assessment and treatment of cardiovascular risk in prediabetes: impaired glucose tolerance and impaired fasting glucose. Am J Cardiol. 2011 Aug 2;108(3 Suppl):3B-24B. doi: 10.1016/j.amjcard.2011.03.013. PMID 21802577
- [Background] Bateman LA, Slentz CA, Willis LH, Shields AT, Piner LW, Bales CW, Houmard JA, Kraus WE. Comparison of aerobic versus resistance exercise training effects on metabolic syndrome (from the Studies of a Targeted Risk Reduction Intervention Through Defined Exercise - STRRIDE-AT/RT). Am J Cardiol. 2011 Sep 15;108(6):838-44. doi: 10.1016/j.amjcard.2011.04.037. Epub 2011 Jul 7. PMID 21741606
- [Background] Malin SK, Nightingale J, Choi SE, Chipkin SR, Braun B. Metformin modifies the exercise training effects on risk factors for cardiovascular disease in impaired glucose tolerant adults. Obesity (Silver Spring). 2013 Jan;21(1):93-100. doi: 10.1002/oby.20235. PMID 23505172
- [Background] Malin SK, Niemi N, Solomon TP, Haus JM, Kelly KR, Filion J, Rocco M, Kashyap SR, Barkoukis H, Kirwan JP. Exercise training with weight loss and either a high- or low-glycemic index diet reduces metabolic syndrome severity in older adults. Ann Nutr Metab. 2012;61(2):135-41. doi: 10.1159/000342084. PMID 23036993
- [Background] Potteiger JA, Claytor RP, Hulver MW, Hughes MR, Carper MJ, Richmond S, Thyfault JP. Resistance exercise and aerobic exercise when paired with dietary energy restriction both reduce the clinical components of metabolic syndrome in previously physically inactive males. Eur J Appl Physiol. 2012 Jun;112(6):2035-44. doi: 10.1007/s00421-011-2174-y. Epub 2011 Sep 23. PMID 21947428
- [Background] Mestek ML, Westby CM, Van Guilder GP, Greiner JJ, Stauffer BL, DeSouza CA. Regular aerobic exercise, without weight loss, improves endothelium-dependent vasodilation in overweight and obese adults. Obesity (Silver Spring). 2010 Aug;18(8):1667-9. doi: 10.1038/oby.2009.467. Epub 2010 Jan 7. PMID 20057377
- [Background] Phillips SA, Mahmoud AM, Brown MD, Haus JM. Exercise interventions and peripheral arterial function: implications for cardio-metabolic disease. Prog Cardiovasc Dis. 2015 Mar-Apr;57(5):521-34. doi: 10.1016/j.pcad.2014.12.005. Epub 2014 Dec 18. PMID 25529367
- [Background] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913
- [Background] Malin SK, Gerber R, Chipkin SR, Braun B. Independent and combined effects of exercise training and metformin on insulin sensitivity in individuals with prediabetes. Diabetes Care. 2012 Jan;35(1):131-6. doi: 10.2337/dc11-0925. Epub 2011 Oct 31. PMID 22040838
- [Background] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Nedeljkovic ZS, Menzoian JO, Vita JA. Predictive value of noninvasively determined endothelial dysfunction for long-term cardiovascular events in patients with peripheral vascular disease. J Am Coll Cardiol. 2003 May 21;41(10):1769-75. doi: 10.1016/s0735-1097(03)00333-4. PMID 12767663
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Eggleston EM, Jahn LA, Barrett EJ. Early microvascular recruitment modulates subsequent insulin-mediated skeletal muscle glucose metabolism during lipid infusion. Diabetes Care. 2013 Jan;36(1):104-10. doi: 10.2337/dc11-2399. Epub 2012 Sep 6. PMID 22961574
- [Background] Liu Z, Liu J, Jahn LA, Fowler DE, Barrett EJ. Infusing lipid raises plasma free fatty acids and induces insulin resistance in muscle microvasculature. J Clin Endocrinol Metab. 2009 Sep;94(9):3543-9. doi: 10.1210/jc.2009-0027. Epub 2009 Jun 30. PMID 19567533
- [Background] Vincent MA, Clerk LH, Lindner JR, Price WJ, Jahn LA, Leong-Poi H, Barrett EJ. Mixed meal and light exercise each recruit muscle capillaries in healthy humans. Am J Physiol Endocrinol Metab. 2006 Jun;290(6):E1191-7. doi: 10.1152/ajpendo.00497.2005. PMID 16682488
- [Background] Barrett EJ, Wang H, Upchurch CT, Liu Z. Insulin regulates its own delivery to skeletal muscle by feed-forward actions on the vasculature. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E252-63. doi: 10.1152/ajpendo.00186.2011. Epub 2011 May 24. PMID 21610226
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702
- [Background] Keske MA, Clerk LH, Price WJ, Jahn LA, Barrett EJ. Obesity blunts microvascular recruitment in human forearm muscle after a mixed meal. Diabetes Care. 2009 Sep;32(9):1672-7. doi: 10.2337/dc09-0206. Epub 2009 Jun 1. PMID 19487636
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Anderson TJ, Charbonneau F, Title LM, Buithieu J, Rose MS, Conradson H, Hildebrand K, Fung M, Verma S, Lonn EM. Microvascular function predicts cardiovascular events in primary prevention: long-term results from the Firefighters and Their Endothelium (FATE) study. Circulation. 2011 Jan 18;123(2):163-9. doi: 10.1161/CIRCULATIONAHA.110.953653. Epub 2011 Jan 3. PMID 21200002
- [Background] Cruickshank K, Riste L, Anderson SG, Wright JS, Dunn G, Gosling RG. Aortic pulse-wave velocity and its relationship to mortality in diabetes and glucose intolerance: an integrated index of vascular function? Circulation. 2002 Oct 15;106(16):2085-90. doi: 10.1161/01.cir.0000033824.02722.f7. PMID 12379578
- [Background] Donley DA, Fournier SB, Reger BL, DeVallance E, Bonner DE, Olfert IM, Frisbee JC, Chantler PD. Aerobic exercise training reduces arterial stiffness in metabolic syndrome. J Appl Physiol (1985). 2014 Jun 1;116(11):1396-404. doi: 10.1152/japplphysiol.00151.2014. Epub 2014 Apr 17. PMID 24744384
- [Background] Green DJ, Eijsvogels T, Bouts YM, Maiorana AJ, Naylor LH, Scholten RR, Spaanderman ME, Pugh CJ, Sprung VS, Schreuder T, Jones H, Cable T, Hopman MT, Thijssen DH. Exercise training and artery function in humans: nonresponse and its relationship to cardiovascular risk factors. J Appl Physiol (1985). 2014 Aug 15;117(4):345-52. doi: 10.1152/japplphysiol.00354.2014. Epub 2014 Jun 19. PMID 24947027
- [Background] Swift DL, Weltman JY, Patrie JT, Saliba SA, Gaesser GA, Barrett EJ, Weltman A. Predictors of improvement in endothelial function after exercise training in a diverse sample of postmenopausal women. J Womens Health (Larchmt). 2014 Mar;23(3):260-6. doi: 10.1089/jwh.2013.4420. Epub 2013 Dec 3. PMID 24299160
- [Background] Mather KJ, Verma S, Anderson TJ. Improved endothelial function with metformin in type 2 diabetes mellitus. J Am Coll Cardiol. 2001 Apr;37(5):1344-50. doi: 10.1016/s0735-1097(01)01129-9. PMID 11300445
- [Background] Vitale C, Mercuro G, Cornoldi A, Fini M, Volterrani M, Rosano GM. Metformin improves endothelial function in patients with metabolic syndrome. J Intern Med. 2005 Sep;258(3):250-6. doi: 10.1111/j.1365-2796.2005.01531.x. PMID 16115299
- [Background] Patel C, Ghanim H, Ravishankar S, Sia CL, Viswanathan P, Mohanty P, Dandona P. Prolonged reactive oxygen species generation and nuclear factor-kappaB activation after a high-fat, high-carbohydrate meal in the obese. J Clin Endocrinol Metab. 2007 Nov;92(11):4476-9. doi: 10.1210/jc.2007-0778. Epub 2007 Sep 4. PMID 17785362
- [Background] Malin SK, Braun B. Impact of Metformin on Exercise-Induced Metabolic Adaptations to Lower Type 2 Diabetes Risk. Exerc Sport Sci Rev. 2016 Jan;44(1):4-11. doi: 10.1249/JES.0000000000000070. PMID 26583801
- [Background] Selvin E, Bolen S, Yeh HC, Wiley C, Wilson LM, Marinopoulos SS, Feldman L, Vassy J, Wilson R, Bass EB, Brancati FL. Cardiovascular outcomes in trials of oral diabetes medications: a systematic review. Arch Intern Med. 2008 Oct 27;168(19):2070-80. doi: 10.1001/archinte.168.19.2070. PMID 18955635
- [Derived] Malin SK, Remchak ME, Heiston EM, Fabris C, Shah AM. Pancreatic beta-cell Function is Higher in Morning Versus Intermediate Chronotypes With Obesity. Obes Sci Pract. 2025 Feb 26;11(2):e70064. doi: 10.1002/osp4.70064. eCollection 2025 Apr. PMID 40018087
- [Derived] Ragland TJ, Heiston EM, Ballantyne A, Stewart NR, La Salvia S, Musante L, Luse MA, Isakson BE, Erdbrugger U, Malin SK. Extracellular vesicles and insulin-mediated vascular function in metabolic syndrome. Physiol Rep. 2023 Jan;11(1):e15530. doi: 10.14814/phy2.15530. PMID 36597186
- [Derived] Remchak ME, Heiston EM, Ballantyne A, Dotson BL, Stewart NR, Spaeth AM, Malin SK. Insulin Sensitivity and Metabolic Flexibility Parallel Plasma TCA Levels in Early Chronotype With Metabolic Syndrome. J Clin Endocrinol Metab. 2022 Jul 14;107(8):e3487-e3496. doi: 10.1210/clinem/dgac233. PMID 35429387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Started | 22 | 21 | 24 | 24
Completed | 16 | 18 | 20 | 18
Not Completed | 6 | 3 | 4 | 6
Not completed — COVID-19 | 3 | 2 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin | Total
Number analyzed (Participants) | 22 | 21 | 24 | 24 | 91
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.5 [50.3 to 63.0] | 54.0 [49.0 to 60.0] | 56.0 [49.8 to 60.0] | 56.0 [49.0 to 64.3] | 56.0 [49.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 19 | 18 | 71
  Male | 5 | 4 | 5 | 6 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 21 | 24 | 21 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 19 | 18 | 23 | 16 | 76
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 31.3 [29.3 to 37.7] | 33.8 [32.6 to 38.8] | 35.3 [32.2 to 38.8] | 36.0 [31.0 to 38.9] | 34.8 [30.9 to 38.8]
VO2peak [Median (Inter-Quartile Range); unit: ml/kg/min] | 22.6 [20.2 to 24.2] | 23.0 [21.2 to 25.3] | 22.9 [20.3 to 26.4] | 21.1 [18.4 to 23.4] | 22.5 [19.7 to 25.1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Unscaled Flow Mediated Dilation (FMD) of the Brachial Artery
Description: Endothelial function assessed as a percentage change in brachial artery diameter from baseline to deflation (5 minutes after artery occlusion by blood pressure cuff inflation). Delta = Week 16 - Week 0. Higher values and positive change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: Percent change in diameters
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 12 | 11 | 16 | 9
Percent change in diameters | -0.45 [-3.47 to 2.56] | 0.76 [-4.17 to 5.70] | 3.50 [0.65 to 6.46] | 5.28 [0.67 to 9.88]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention 0 min unscaled FMD change, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.045, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.017; Linear ANCOVA model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 3.53, 95% CI 2-sided [0.08 to 6.99]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.507, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.050; ANCOVA linear model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-2.42 to 4.73]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.014, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.008; ANCOVA linear model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 4.98, 95% CI 2-sided [1.14 to 8.83]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.237, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.033; ANCOVA linear model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 2.38, 95% CI 2-sided [-1.66 to 6.42]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.486, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.042; ANCOVA linear model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 1.45, 95% CI 2-sided [-2.80 to 5.70]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.081, ANCOVA — Benjamini and Hochberg method was used to decrease the false discovery rate with an overall error rate of 0.05. The B&H P-value threshold for this comparison was 0.025; ANCOVA linear model adjusted for pre-intervention FMD; Mean Difference (Final Values) = 3.83, 95% CI 2-sided [-0.53 to 8.19]

2. Secondary Outcome: Change in Metabolic Insulin Sensitivity. Glucose Infusion Rate Normalized to Steady-State Insulin (GIR).
Description: The glucose infusion rate (mg/kg/min) divided by steady-state insulin (uU/mL) during a 120 minute euglycemic-hyperinsulinemic clamp provides an index of metabolic insulin sensitivity. Delta = Week 16 - Week 0. Higher values and positive change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: (mg/kg/min)/(uU/mL)
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 14 | 16 | 19 | 14
(mg/kg/min)/(uU/mL) | 0.0012 [-0.0131 to 0.0155] | 0.011 [0.0047 to 0.0173] | 0.0086 [-0.0011 to 0.0182] | 0.0053 [-0.0051 to 0.0158]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention GIR, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.373, ANCOVA — [p-value comment as in outcome 1, analysis 6]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = 0.0073, 95% CI 2-sided [-0.0093 to 0.0240]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.198, ANCOVA — [p-value comment as in outcome 1, analysis 3]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = 0.0097, 95% CI 2-sided [-0.0055 to 0.0250]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.622, ANCOVA — [p-value comment as in outcome 1, analysis 4]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = 0.0041, 95% CI 2-sided [-0.0129 to 0.0211]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.666, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = -0.0024, 95% CI 2-sided [-0.0136 to 0.0088]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.634, ANCOVA — [p-value comment as in outcome 1, analysis 5]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = -0.0032, 95% CI 2-sided [-0.0169 to 0.0104]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.336, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA linear model adjusted for pre-intervention GIR; Mean Difference (Final Values) = -0.0056, 95% CI 2-sided [-0.0174 to 0.0062]

3. Secondary Outcome: Change in Fasting Augmentation Index
Description: Measure of Arterial Stiffness calculated by dividing the augmentation pressure by the pulse pressure, then multiplying by 100 and normalizing to a heart rate of 75 bpm (AIx75). Delta = Week 16 - Week 0. Lower values and negative change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: Percent of pulse pressure
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 15 | 17 | 20 | 15
Percent of pulse pressure | -1.33 [-7.84 to 5.17] | -4.65 [-9.35 to 0.06] | 0.00 [-4.81 to 4.81] | -1.20 [-4.50 to 2.10]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention AIx75 change, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.671, ANCOVA — [p-value comment as in outcome 1, analysis 5]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [-5.68 to 8.69]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.170, ANCOVA — [p-value comment as in outcome 1, analysis 6]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = -4.82, 95% CI 2-sided [-11.84 to 2.19]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.839, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-7.29 to 5.97]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.024, ANCOVA — [p-value comment as in outcome 1, analysis 3]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = 6.33, 95% CI 2-sided [0.86 to 11.80]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.385, ANCOVA — [p-value comment as in outcome 1, analysis 4]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-7.16 to 2.83]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.080, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA linear model adjusted for pre-intervention AIx75; Mean Difference (Final Values) = 4.17, 95% CI 2-sided [-0.53 to 8.86]

4. Secondary Outcome: Change in Insulin-stimulated Microvascular Blood Flow (MBF) of the Forearm.
Description: Product of microvascular blood volume (VI; video intensity units) and microvascular flow velocity (sec^-1). Insulin-stimulated microvascular blood flow is the change during a 120 minute euglycemic-hyperinsulinemic clamp (120-0 minutes). Delta = Week 16 - Week 0. Higher values and positive change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: VI * sec^-1
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 10 | 7 | 15 | 7
VI * sec^-1 | 0.027 [-0.003 to 0.056] | 0.041 [-0.037 to 0.119] | -0.026 [-0.059 to 0.007] | -0.065 [-0.128 to -0.001]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention MBF change, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.088, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = -0.032, 95% CI 2-sided [-0.069 to 0.005]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.960, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.059 to 0.062]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.075, ANCOVA — [p-value comment as in outcome 1, analysis 3]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = -0.052, 95% CI 2-sided [-0.109 to 0.006]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.258, ANCOVA — [p-value comment as in outcome 1, analysis 4]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = -0.033, 95% CI 2-sided [-0.094 to 0.028]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.443, ANCOVA — [p-value comment as in outcome 1, analysis 5]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = -0.020, 95% CI 2-sided [-0.075 to 0.035]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.144, ANCOVA — [p-value comment as in outcome 1, analysis 6]; ANCOVA linear model adjusted for pre-intervention MBF; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-0.126 to 0.020]

5. Secondary Outcome: Change in Insulin-stimulated Microvascular Flow Velocity (MFV) of the Forearm.
Description: Replenishment curves of the forearm flexor muscle acquired during steady-state infusion of Definity microbubbles. Insulin-stimulated microvascular flow velocity is the change during a 120 minute euglycemic-hyperinsulinemic clamp (120-0 minutes). Delta = Week 16 - Week 0. Higher values and positive change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: sec^-1
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 10 | 7 | 15 | 7
sec^-1 | 0.006 [-0.004 to 0.015] | 0.009 [-0.013 to 0.032] | -0.007 [-0.017 to 0.003] | -0.018 [-0.035 to -0.001]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention MFV change, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.147, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.017 to 0.003]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.943, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.016 to 0.017]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.108, ANCOVA — [p-value comment as in outcome 1, analysis 3]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.027 to 0.003]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.319, ANCOVA — [p-value comment as in outcome 1, analysis 4]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.024 to 0.009]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.496, ANCOVA — [p-value comment as in outcome 1, analysis 5]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.019 to 0.010]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.187, ANCOVA — [p-value comment as in outcome 1, analysis 6]; ANCOVA linear model adjusted for pre-intervention MFV; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.031 to 0.007]

6. Secondary Outcome: Change in Insulin-stimulated Microvascular Blood Volume (MBV) of the Forearm.
Description: Replenishment curves of the forearm flexor muscle acquired during steady-state infusion of Definity microbubbles. Insulin-stimulated microvascular blood volume is the change during a 120 minute euglycemic-hyperinsulinemic clamp (120-0 minutes). Delta = Week 16 - Week 0. Higher values and positive change scores following the intervention indicate a better outcome.
Time Frame: 0 and 16 weeks
Population: Analysis includes only individuals that had both pre and post data.
Measure: Mean (95% Confidence Interval); unit: Video Intensity Units (VI)
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
Number analyzed (Participants) | 10 | 7 | 15 | 7
Video Intensity Units (VI) | 0.188 [-0.015 to 0.392] | 0.433 [-0.229 to 1.096] | -0.257 [-0.520 to 0.006] | -0.510 [-1.046 to 0.026]
Statistical Analysis 1: Comparison: LoEx With Placebo vs LoEx With Metformin; Intention to treat Full Maximum Likelihood based comparisons of baseline covariate adjusted pre- to post-intervention MBV change, where the difference is between treatment combination #2 and treatment combination #1 (i.e. treatment combination # 2 - treatment combination #1); Test type: Superiority; p = 0.086, ANCOVA — [p-value comment as in outcome 1, analysis 3]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = -0.230, 95% CI 2-sided [-0.495 to 0.035]
Statistical Analysis 2: Comparison: LoEx With Placebo vs HiEx With Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.608, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [-0.354 to 0.574]
Statistical Analysis 3: Comparison: LoEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.110, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = -0.344, 95% CI 2-sided [-0.779 to 0.090]
Statistical Analysis 4: Comparison: HiEx With Placebo vs LoEx With Metformin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.145, ANCOVA — [p-value comment as in outcome 1, analysis 4]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = -0.340, 95% CI 2-sided [-0.818 to 0.137]
Statistical Analysis 5: Comparison: LoEx With Metformin vs HiEx With Metformin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.565, ANCOVA — [p-value comment as in outcome 1, analysis 5]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = -0.114, 95% CI 2-sided [-0.538 to 0.309]
Statistical Analysis 6: Comparison: HiEx With Placebo vs HiEx With Metformin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.110, ANCOVA — [p-value comment as in outcome 1, analysis 6]; ANCOVA linear model adjusted for pre-intervention MBV; Mean Difference (Final Values) = -0.454, 95% CI 2-sided [-1.025 to 0.116]

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the first dose of double-blind study medication and within 14 days after the last dose of double-blind study medication, an average of 18 weeks.
Description: Any event reported by the participant or observed by the study staff was was documented and reported to the Institutional Review Board, irrespective of the relation to the research study. Adverse events were collected in a non-systematic method by which participants reported events or in response to to open-ended questions, which occurred once every week for 16 weeks.
Arm/Group | LoEx With Placebo | HiEx With Placebo | LoEx With Metformin | HiEx With Metformin
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LoEx With Placebo (N=22) | HiEx With Placebo (N=21) | LoEx With Metformin (N=24) | HiEx With Metformin (N=24)
Gastrointestinal Distress (Gastrointestinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to unforeseen technical issues with the vascular imaging files, we were regrettably unable to analyze the endothelial function data (FMD) for a majority of participants who had been randomized to HiEx with Metformin group, as well as others in the remaining 3 treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03355469/Prot_SAP_002.pdf
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03355469/ICF_003.pdf